CLINICAL TRIAL: NCT01396785
Title: A Randomized, Multi-Center, Double-Blind, Vehicle-Controlled Study Evaluating the Efficacy and Safety of Product 33525 in Subjects With Tinea Pedis
Brief Title: Topical Antifungal Treatment for Tinea Pedis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medicis Global Service Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MP-1000-02
Record Dates: First submitted 2011-07-15; First posted 2011-07-19 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: Tinea Pedis
Keywords: Tinea Pedis; Antifungal
MeSH Terms: conditions — Tinea Pedis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental): Product 33525
  Interventions: Drug: 33525
- Placebo (Placebo Comparator): Product 33525 Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 33525 — Daily for 14 days
  Arms: Active
Drug: Placebo — Daily for 14 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if a topical antifungal cream is safe and effective for the treatment of tinea pedis.

ELIGIBILITY:
Inclusion Criteria:

* Moderate erythema, moderate scaling, and mild pruritus

Exclusion Criteria:

* Pregnancy and allergies

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2011-07; Primary Completion 2012-01 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Proportion of patients achieving complete clearance | Day 42
  Signs and Symptoms Severity Score and negative Potassium Hydroxide (KOH) and Culture

SECONDARY OUTCOMES:
Proportion of patients achieving effective treatment | Day 42
  Clinical Cure and Mycologic Cure

CONTACTS AND LOCATIONS:
Overall Officials: Ron Staugaard, Study Director — Medicis Pharmaceutical
Locations (10):
- United States (9):
  - Los Angeles, California
  - Paramus, New Jersey
  - Albuquerque, New Mexico
  - Hershey, Pennsylvania
  - Austin, Texas
  - College Station, Texas
  - Plano, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
- Cidra, Puerto Rico